CLINICAL TRIAL: NCT02966366
Title: Tinnitus Treatment With Cochlear Implant in Single Sided Deafness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIC_02
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Single Sided Deafness; Tinnitus; Cochlear Implant
MeSH Terms: conditions — Tinnitus | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear implantation (Experimental): Evaluation of tinnitus before and after cochlear implantation
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant

SUMMARY:
Recent studies have reported successful reduction of tinnitus after cochlear implantation (CI) in most CI users, but the mechanisms of reduction and the amount of improvement is not fully understood. Especially, the relative role of peripheral and central auditory pathways is not clearly known. This study assessed the effect of CI electrical stimulation on tinnitus in subjects with unilateral tinnitus related to a single-sided deafness (SSD), and relative contributions of peripheral and central auditory pathways in tinnitus reduction.

DETAILED DESCRIPTION:
Introduction: Continuous surgical, technological and audiological advances are responsible for the ever improvement of outcomes obtained through cochlear implants (CI) over the last decades. These positive observations have progressively led to the cautious extension of CI indications including patients with single-sided deafness (SSD). SSD patients are characterized by the loss of functional hearing in one ear, causing an impairment of binaural hearing abilities, with important difficulties for sound localization and speech in noise comprehension. These patients also often present invalidating tinnitus in the deaf ear, worsening both their psychological and audiological conditions. Recent studies have reported successful reduction of tinnitus intensity after cochlear implantation. However, most studies included a very limited number of participants and tinnitus evaluation tools. The impact of CI speech perception abilities in SSD is still under debate.

Objective: This study aims to assess the effect of CI electrical stimulation on tinnitus, speech-in-noise and speech-in-quiet abilities in a group of 30 SSD patients.

Methods: After cochlear implantation, patients are stimulated using continuous white noise stimulation in the first month period and thereafter using a conventional stimulation. This was done to investigate the effects of non-meaningful, and therefore only peripheral, stimulation. Outcomes were monitored at 1, 3, 6 and 12 months of CI use. Tinnitus loudness and annoyance were measured with a Visual Analog Scale and tinnitus distress and quality of life were evaluated with tinnitus questionnaires (THI, TRQ and STSS). Speech in noise comprehension was assessed in three different spatial listening configurations and speech in quiet was evaluated through direct connection with the speech processor.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Profound to total single sided deafness with associated tinnitus
* Normal or near-normal hearing on contralateral ear
* Tinnitus evaluated by THI ≥ 58 and VAS on annoyance ≥8
* Failure of usual tinnitus treatments
* Duration of tinnitus between 1 and 15 years
* Normal vestibular function of contralateral ear
* Native of fluent French speaker

Exclusion Criteria:

* No Social security affiliation
* Retrocochlear pathology (vestibular schwannoma, severe central auditory processing disorder)
* Cochlear ossification
* Middle ear pathology
* Tinnitus not related to deafness
* Depression with BDI (Beck Depression Inventory) > 16 or unfavorable advice from psychologist/ psychiatrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Change for Visual Analog Scale (VAS) on Intensity and annoyance between pre and post implantation | Change from pre-implantation Visual Analog Scale (VAS) scores on intensity and annoyance at 1 month after white noise stimulation, 1, 3, 6 and 12 months after conventional stimulation
change for THI Tinnitus Handicap Inventory scale between pre and post implantation | Change from pre-implantation scores on Tinnitus Handicap Inventory Scale (THI scale) at 1 month after white noise stimulation, 1, 3, 6 and 12 months after conventional stimulation
Change for TRQ Tinnitus Reaction Questionnaire between pre and post implantation | Change from pre-implantation scores on Tinnitus Reaction Questionnaire (TRQ) at 1 month after white noise stimulation, 1, 3, 6 and 12 months after conventional stimulation
Change for STSS Subjective Tinnitus Severity Scale between pre and post implantation | Change from pre-implantation scores on Subjective Tinnitus Severity Scale (STSS) at 1 month after white noise stimulation, 1, 3, 6 and 12 months after conventional stimulation

SECONDARY OUTCOMES:
Speech in noise intelligibility | Before cochlear implantation, 6 and 12 after conventional stimulation
  Comparison of speech intelligibility in noise with and without the speech processor, when measured in free field, with the normal hearing ear unplugged. Performance (% of words correctly repeated) is measured:
  * With two level of noise (Speech to Noise Ratio of -3dB and +5 dB)
  * In three different spatial configurations: (S0N0: signal and noise coming from the front; S0NIC: Signal coming from the front and noise coming from the implanted side; SICN0: Signal coming from the implanted side and noise coming from the front.
Speech in quiet intelligibility with cochlear implant only | 6 and 12 after conventional stimulation
  Speech intelligibility for speech in quiet with the cochlear implant only (speech signals presented through direct connection).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Gnansia, Dr, Study Director — Oticon Medical; Bruno Frachet, Pr, Principal Investigator — Hôpital Rothschild
Locations (6):
- France (6):
  - CHRU Lille Hôpital Roger Salengro, Lille
  - CHU Lyon Hôpital Edouard Herriot, Lyon
  - Hôpital la Pitié Salpêtrièr, Paris
  - Hôpital Rothschild, Paris
  - CHU Rennes Pontchaillou, Rennes
  - CHU Tours Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No